CLINICAL TRIAL: NCT04216758
Title: An Exploratory Clinical Trial of Nab-Paclitaxel and Gemcitabine Compared With Gemcitabine and Tegafur in Adjuvant Chemotherapy After Radical Resection of Pancreatic Cancer
Brief Title: Nab-P and Gem Compared With Gem and Tegafur in Adjuvant Chemotherapy After Radical Resection of Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Principal Investigator, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-23
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Stage IA Pancreatic Adenocarcinoma; Stage IB Pancreatic Adenocarcinoma; Stage IIA Pancreatic Adenocarcinoma; Stage IIB Pancreatic Adenocarcinoma
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Tegafur

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nab-paclitaxel + gemcitabine (Experimental): nab-paclitaxel at 100 mg/m^2 on days 1, 8, and 15; gemcitabine at 1000 mg/m^2 on days 1, 8, and 15
  Interventions: Drug: nab-paclitaxel; Drug: Gemcitabine
- tegafur + gemcitabine (Experimental): gemcitabine at 1000 mg/m^2 on days 1, 8, and 15; tegafur: Body surface area < 1.25 m^2, 60 mg/d; Body surface area ≥ 1.25 m^2 to < 1.5 m^2, 80 mg/d; Body surface area ≥ 1.5 m^2, 100 mg/d; Oral (po), Bid, D1-21
  Interventions: Drug: Gemcitabine; Drug: tegafur

INTERVENTIONS:
Drug: nab-paclitaxel — Patients firstly receive nab-paclitaxel 100 mg/m^2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks for up to 6 circles in the absence of disease recurrence or unacceptable toxicity.
  Other Names: Abraxane
  Arms: nab-paclitaxel + gemcitabine
Drug: Gemcitabine — Patients receive gemcitabine 1000 mg/m^2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks for up to 6 circles in the absence of disease recurrence or unacceptable toxicity.
  Other Names: Gemzar
Drug: tegafur — Patients secondly receive tegafur Body surface area < 1.25 m^2, 60 mg/d;Body surface area ≥ 1.25 m^2 to < 1.5 m^2, 80 mg/d;Body surface area ≥ 1.5 m^2, 100 mg/d (po) on days 1-21 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks for up to 6 circles in the absence of disease recurrence or unacceptable toxicity.
  Arms: tegafur + gemcitabine

SUMMARY:
Treatment, Prospective, Assignment, Open Label, Single-center, Non-randomized Study An exploratory clinical trial of comparison of Nab-Paclitaxel combined with Gemcitabine and Gemcitabine combined with Tegafur for adjuvant chemotherapy after radical resection of pancreatic cancer

DETAILED DESCRIPTION:
Pancreatic cancer has an extremely poor prognosis with a 5-year survival rate of less than 5%. About 25% of patients have the opportunity for radically surgical resection when diagnosis. However, the recurrence rate is up to 85% within 2 years. Data from clinical trials indicated that gemcitabine-based adjuvant chemotherapy reduced recurrence and enhanced overall survival for patients who have undergone surgery to remove their tumor. Nab-paclitaxel could significantly increase the concentration of gemcitabine in the tumor; recent studies showed that nab-paclitaxel plus gemcitabine significantly improved progression-free survival and overall survival of metastatic pancreatic cancer patients. A study in Japan and Taiwan compared the efficacy of gemcitabine in combination with tegafur in patients with locally advanced or metastatic pancreatic cancer. The median progression-free survival was significantly better in the gemcitabine combined with the tegafur group than in the gemcitabine group. The present study is intended to observe the effect of albumin paclitaxel combined with gemcitabine and tegafur combined with gemcitabine on recurrence-free survival in patients with pancreatic adenocarcinoma undergoing radical resection.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment
* Age ≥18 years and ≤ 80 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Pathologically confirmed after R0 resection of pancreatic adenocarcinoma.
* The expected survival after surgery ≥ 6 months
* No serious blood system, heart, lung function abnormalities and immune defects (refer to the respective standards)
* White blood cell (WBC) ≥ 3 × 109/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelets (PLT) ≥ 100 × 109/L; Hemoglobin (Hgb)≥ 9 g/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤ 2.5 × institutional upper limit of normal (ULN); Total bilirubin (TBIL) ≤ ULN; Creatinine (CRE) ≤ 1.5 × ULN
* Prothrombin time (PT) and international normalized ratio (INR) ≤ 1.5 ×ULN
* Baseline (postoperative) abdominal pelvic CT (plain scan + enhancement) and chest CT scan without tumor lesions;
* No serious adverse events (fatal or life-threatening, persistent or significant loss of function or disability, requiring hospitalization or prolonged hospital stay) within 4-12 weeks after surgery;
* Comply with research visit plans and other program requirements.

Exclusion Criteria:

* with other systemic malignancies
* Patients who have received any form of anti-tumor therapy before surgery, including chemotherapy, radiotherapy, interventional chemoembolization, radiofrequency ablation, and molecular targeted therapy
* used any other study drug within 5 weeks prior to enrollment;
* Patients with central nervous system diseases, mental illness, unstable angina pectoris, congestive heart failure, severe arrhythmia and other serious diseases that cannot be controlled
* Uncontrolled infection, hemorrhage, pancreatic leakage, bile leakage, or other postoperative complications during baseline examination; acute and chronic metabolic acidosis (including ketoacidosis, lactic acidosis) failed to be corrected;
* History of allergic reactions attributed to compounds of similar chemical or biological composition to nab-paclitaxel or gemcitabine or tegafur
* Pregnant or nursing women
* Any condition that may compromise patient safety or study data integrity, including serious medical risk factors, medical conditions, and laboratory abnormalities;
* Patients may leave the observation for 7 days or more during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) | From date of the first day after surgery until the date of the recurrence of the disease (local recurrence and/or distant metastasis) or death from any cause,whichever came first, assessed up to 20 months
  To evaluate the therapeutic efficacy of comparison of Nab-Paclitaxel combined with Gemcitabine and Gemcitabine combined with Tegafur chemotherapy in terms of recurrence-free survival in patients with pancreatic cancer after curative resection. Computed tomography (CT) scan

SECONDARY OUTCOMES:
Overall survival (OS) | From date of enrollment (after curative resection) until the date of death from any cause, assessed one month during therapy and 3 months thereafter
  To evaluate the overall survival of patients (after curative resection) treated with this regimen. Outpatient visit, phone interview
Quality of life (Qol) | One month during therapy and 3 months thereafter
  To evaluate the quality of life score of patients (after curative resection) treated with this regimen. Outpatient visit, phone interview
Number of grade 3 and 4 toxicities according to NCI CTCAE version 4.0 | One week during therapy and 3 months thereafter
  To evaluate the occurrence of grade 3 and 4 toxicities according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE; version 4.0) in patients treated with this regimen. The toxicity profile includes but not limits neutropenia, thrombocytopenia, peripheral neuropathy, hypoglycemia, metabolic acidosis (acute or chronic, including ketoacidosis), which will be summarized as the percentage of patients by type and grade according to treatment group. Outpatient visit, laboratory findings
CA199 level after curative resection | One month during therapy and 3 months thereafter
  To evaluate the CA199 level of patients (after curative resection) treated with this regimen. Outpatient visit, laboratory findings

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Yu, M.D Ph.D, Principal Investigator — Fudan University
Locations (1):
- Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University; 270 Dong An Road, Shanghai 200032, China, Shanghai, China

IPD SHARING:
Plan to Share IPD: No